CLINICAL TRIAL: NCT01155219
Title: Safety and Efficacy Assessment of Geltim LP® 1 mg/g (Unpreserved Timolol Gel - TG1030) in Ocular Hypertensive or Glaucomatous Patients Stabilized by Xalatan® With Ocular Intolerance Signs.
Brief Title: Safety, Efficacy Assessment of Geltim LP® 1 mg/g in Ocular Hypertensive or Glaucomatous Patients.
Acronym: T1030
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LTG1030-PIV-12/07
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Results first posted 2014-10-29 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2010-07

CONDITIONS: Glaucoma
Keywords: Bilateral Glaucoma; Bilateral ocular hypertension; Bilateral primary open angle glaucoma; Bilateral ocular hypertension already treated and controlled by mono-therapy of Xalatan® (1drop per day); With local intolerance signs in at least one eye
MeSH Terms: conditions — Glaucoma | interventions — Latanoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Geltim LP® (Experimental): Geltim LP® 1 mg/g (0.1 % timolol maleate, without preservative) packaged in single-dose containers (unidoses); one drop in the conjunctival sac of each eye in the morning (84 days).
  Interventions: Drug: Geltim LP 1 mg/g
- Xalatan® (Active Comparator): Xalatan® (Latanaprost) aqueous eye drop (one drop in the conjunctival sac of each eye in the evening during 84 days.
  Interventions: Drug: Xalatan

INTERVENTIONS:
Drug: Geltim LP 1 mg/g — one drop in the conjunctival sac of each eye in the morning (84 days).
  Arms: Geltim LP®
Drug: Xalatan — one drop in the conjunctival sac of each eye in the morning (84 days).
  Arms: Xalatan®

SUMMARY:
This phase IV study aims to assess the safety and the efficacy in intra ocular pressure of Geltim LP® 1 mg/g (0.1% unpreserved timolol maleate gel) in glaucomatous patients initially treated and stabilised by monotherapy of Xalatan® with ocular objective signs of intolerance to prostaglandin eye drops.

DETAILED DESCRIPTION:
The primary objectives are to compare the safety and the efficacy of Geltim LP® 1mg/g eye drops versus Xalatan® eye drops with respect to:

The assessment of the ocular tolerance:

* Ocular symptoms
* Objective ocular signs.

The maintain of the IOP efficient lowering effect. Comparison between the 2 study products of the mean basal IOP after a 12 weeks treatment period (84 days ±7).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Association of the 4 following criteria:

  1. - Bilateral primary open angle glaucoma or bilateral ocular hypertension already treated and controlled by mono-therapy of Xalatan® (1drop per day),
  2. - With local intolerance signs.

Exclusion Criteria:

* Presence of severe objective ocular sign.
* Any ocular hypertension other than primary ocular hypertension or primary chronic open angle glaucoma (such as congenital, angle closure glaucoma, secondary glaucoma).
* Absolute defect in the ten degrees central point of the visual field.
* Best far corrected visual acuity ≤ 1/10.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clermont-Ferrand, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Geltim LP® | Xalatan®
Started | 77 | 73
Completed | 73 | 70
Not Completed | 4 | 3
Not completed — Adverse Event | 3 | 1
Not completed — non-medical reason | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Geltim LP® | Xalatan® | Total
Number analyzed (Participants) | 77 | 73 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.94 (11.79) | 64.86 (11.62) | 65.41 (11.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 50 | 99
  Male | 28 | 23 | 51
Region of Enrollment [Number; unit: participants]
  France | 77 | 73 | 150

OUTCOME MEASURES:

1. Primary Outcome: Ocular Tolerance
Description: Response defined as a combination of satisfactory or acceptable effect on IOP and a reduction of at least 20% of the total tolerance score in the worse eye.
Time Frame: Day 84
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Geltim LP® | Xalatan®
Number analyzed (Participants) | 71 | 70
participants | 65 | 34
Statistical Analysis 1: Comparison: Geltim LP® vs Xalatan®; Test type: Superiority or Other; p < 0.001, Fisher Exact

ADVERSE EVENTS:
Groups:
- Geltim LP®: Geltim LP® 1 mg/g (0.1 % unpreserved timolol maleate gel)
  One drop in the conjunctival sac of each eye in the morning
- Xalatan®: Latanoprost
  One drop in the conjunctival sac of each eye in the evening
Arm/Group | Geltim LP® | Xalatan®
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/73
Other Adverse Events (participants affected / at risk) | 0/77 | 0/73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the results of the Trial are the sole and exclusive property of THEA, and cannot be used in whatever form without prior written agreement of THEA.